CLINICAL TRIAL: NCT02241200
Title: A Randomized, 2 Part, 4-treatment, 2-way Cross-over Study in Healthy Volunteers to Compare the Pharmacokinetic and Pharmacodynamic Profiles of 1ug/kg of DA-3880 and EU Sourced ARANESP® (Amgen) After Single Intravenous or Subcutaneous Administration
Brief Title: A Study in Healthy Volunteers to Compare the Profiles of DA-3880 and EU Sourced ARANESP® (Amgen)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA3880_ANE_I
Record Dates: First submitted 2014-08-29; First posted 2014-09-16 (Estimated); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Symptomatic Anemia
MeSH Terms: interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV Administration (Experimental): The iv solutions containing DA-3880 and Aranesp will be indistinguishable in appearance.
  Interventions: Drug: DA3880; Drug: Aranesp
- SC Administration (Experimental): The sc solutions containing DA-3880 and Aranesp will be indistinguishable in appearance.
  Interventions: Drug: DA3880; Drug: Aranesp

INTERVENTIONS:
Drug: DA3880
Drug: Aranesp

SUMMARY:
The main purpose of the study is to determine whether the test product and the reference product are bioequivalent based on the pharmacokinetics after administration of ug/kg as a single intravenous dose and as a single subcutaneous dose of each of the formulations. The study is consisted of randomization, 2 parts, 4 treatments, 2 way cross over.

ELIGIBILITY:
Inclusion Criteria:

1. Gender : male or female
2. Age : 18 - 65 years, inclusive
3. Body Mass Index (BMI) : 18.0 - 30.0 kg/m2, inclusive
4. Weight : 55 - 105 kg, inclusive
5. Female subjects of childbearing potential must be non-pregnant and non-lactating, and have a negative pregnancy test at screening and (each) admission to the clinical research center
6. Females of child-bearing potential, with a fertile male sexual partner, should be willing to use adequate contraception from screening until 90 days after the follow-up visit. Adequate contraception is defined as using hormonal contraceptives or an intrauterine device combined with at least 1 of the following forms of contraception: a diaphragm or cervical cap, or a condom.
7. Males should be willing to use adequate contraception and not donate sperm from first admission to the clinical research center until 90 days after the follow-up visit. Adequate contraception for the male subject and his female partner, is defined as using hormonal contraceptives or an intrauterine device combined with at least 1 of the following forms of contraception: a diaphragm or cervical cap, or a condom.
8. All non-regular medication (including over the counter medication, health supplements, and herbal remedies such as St. John's Wort extract) must have been stopped at least 14 days prior to (the first) admission to the clinical research center. An exception is made for paracetamol (acetaminophen), which is allowed up to admission to the clinical research center. Other exceptions are multivitamins and vitamin C, which are allowed up to 7 days before admission to the clinical research center.
9. All regular non-topical medication must have been stopped at least 30 days prior to (the first) admission the clinical research center. An exception is made for hormonal contraceptives, which may be used throughout the study.
10. Ability and willingness to abstain from alcohol, methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, "powerdrinks"), grapefruit (juice) and tobacco products from 48 h prior to each admission to in the clinical research center
11. Medical history without major pathology as judged by the PI
12. Normal resting supine blood pressure and pulse showing no clinically relevant deviations as judged by the PI.
13. Computerized (12-lead) electrocardiogram (ECG) recording without signs of clinically relevant pathology or showing no clinically relevant deviations as judged by the PI.
14. All values for clinical laboratory tests of blood and urine within the normal range or showing no clinically relevant deviations as judged by the PI. Hb, Hct, RBC count and thrombocytes should not exceed the upper limit of normal. Minor deviations can be accepted at the discretion of the PI
15. Willing and able to sign the ICF

Exclusion Criteria:

1. Evidence of clinically relevant pathology
2. Mental handicap
3. History of relevant drug and/or food allergies, and/or latex allergy
4. Smoking more than 10 cigarettes, 2 cigars or 2 pipes daily; the use of tobacco products in the 48 hours (2 days) prior to each admission to the clinical research center is not allowed.
5. History of alcohol or drug abuse or drug addiction (including soft drugs like cannabis products)
6. Positive drug screen (opiates, methadone, cocaine, amphetamines [including ecstasy], cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants and alcohol)
7. Average intake of more than 24 units of alcohol per week: one unit of alcohol equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits)
8. Consumption of any foods containing poppy seeds within 48 hours (2 days) prior to each admission to the clinical research center as this could cause a false positive drug screen result
9. Positive screen on hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies or anti-HIV 1 and 2 antibodies
10. Participation in a drug study within 60 days prior to the screening visit in the current study. Participation in more than 3 other drug studies (for men) and more than 2 other drug studies (for women) in the 10 months prior to the first drug administration in the current study
11. Donation or loss of more than 100 mL of blood within 60 days prior to the first drug administration. Donation or loss of more than 1.5 liters of blood (for men) / more than 1.0 liters of blood (for women) in the 10 months prior to the first drug administration in the current study.
12. Strenuous exercise within 96 hours (4 days) prior to each admission to the clinical research center.
13. Significant and/or acute illness within 5 days prior to the first drug administration that may impact safety assessments, in the opinion of the PI
14. Vaccination within 30 days prior to entry into the clinical research center or planning a vaccination before the follow-up visit
15. History of a significant respiratory disorder (such as asthma) or significant immune disorder
16. Significant infection within 30 days prior to entry into the clinical research center
17. History of epilepsy; a single febrile convulsion at an age < 6 years is acceptable
18. History of hemoglobinopathy or abnormal Hb in first-degree relatives
19. A previous administration of any erythropoiesis-stimulating agent including EPO or darbepoetin, if known
20. Previous immunoglobulin or iron supplementation within 3 months prior to the screening visit
21. History of hypersensitivity reactions for any EPO, darbepoetin, iron supplements, or excipient of the investigational product

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-08-18 (Actual); Primary Completion 2014-11-29 (Actual); Study Completion 2014-11-29 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of DA-3880 and Aranesp via IV Administration | 6 weeks
  AUC0-t, Cmax, Tmax, t½, AUC0-inf, %AUC of DA-3880 and EU sourced Aranesp® (Amgen) after administration of 1 μg/kg as a single iv dose will be assessed.
Pharmacokinetics of DA-3880 and Aranesp via SC Administration | 6 weeks
  AUC0-t, Cmax, Tmax, t½, AUC0-inf, %AUC of DA-3880 and EU sourced Aranesp® (Amgen) after administration of 1 μg/kg as a single sc dose will be assessed

SECONDARY OUTCOMES:
Pharmacodynamic Variables of DA-3880 and Aranesp | 6 weeks
  AUEC0-t, Emax, Tmax of DA-3880 and EU sourced Aranesp® after administration of 1 μg/kg as a single iv dose and as a single sc dose will be assessed.
Safety and Tolerability Parameters of DA-3880 and Aranesp | 6 weeks
  Adverse events, vital signs, 12-lead ECG, clinical laboratory tests, physical examination, immunogenicity (anti-drug antibodies), local tolerability of DA-3880 and EU sourced Aranesp® after administration of 1 μg/kg as a single iv dose and as a single sc dose will be assessed.
Pharmacodynamic and Pharmacodynamic Variables of IV and SC Administration | 6 weeks
  AUC0-t, Cmax, Tmax, t½, AUC0-inf, %AUC, AUEC0-t, Emax, Tmax of DA-3880 (1 μg/kg) and EU sourced Aranesp® (1 μg/kg) after iv administration with those after sc administration will be assessed.
Safety and Tolerability Parameters of SC and IV Administration | 6 weeks
  Adverse events, vital signs, 12-lead ECG, clinical laboratory tests, physical examination, immunogenicity (anti-drug antibodies), local tolerability of DA-3880 (1 μg/kg) and EU sourced Aranesp® (1 μg/kg) after iv administration with those after sc administration will be compared and assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- PRA, Zuidlaren, Netherlands